CLINICAL TRIAL: NCT04809662
Title: Comparing Immune Responses to Topical Imiquimod
Status: Terminated | Type: Observational
Why Stopped: PI failed to submit the study for continuing review to IRB, failed to respond.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1646493
Record Dates: First submitted 2021-03-04; First posted 2021-03-22 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Actinic Keratoses
Keywords: imiquimod; aldara
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main cohort: This is a split-body study, with patients acting as their own controls between lesional and nonlesional skin. All patients will apply imiquimod.
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Drug: Imiquimod — Patients with a diagnosis of actinic keratosis or warts that would be prescribed imiquimod as standard of care will be asked to apply 2 packets (or 2 full pumps) of imiquimod once daily before bedtime for two weeks and then leave on overnight for ~8 hours.
  (a) A biopsy will be performed at the baseline visit on the pre-treatment skin and the skin where the medication will not be applied. The skin where the medication will not be applied will act as the negative control. A biopsy will then again be performed on day 10 of imiquimod treatment on the treated skin only, where the study drug was applied.
  Other Names: Aldara; Zyclara

SUMMARY:
The study is a basic science research study that is designed to characterize and compare the immune response in individuals who are designated as ABO blood group secretors, meaning they have a functional copy of the FUT2 gene versus those patients who are designated ABO non-secretors after application of topical imiquimod to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 to 85 years of age
* Patients with a diagnosis that will result in treatment with imiquimod as standard of care, specifically actinic keratosis

Exclusion Criteria:

* Younger than 18 years or older than 85 years.
* History of hypersensitivity/ allergic reaction or adverse reaction to imiquimod
* Individuals with a diagnostic biopsy and supportive histology of a cutaneous immune-mediated disease (e.g. psoriasis and mycosis fungoides, etc.) or diseases of the hematopoietic system, liver and the gastrointestinal tract (e.g. aplastic anemia, Crohn's disease, Ulcerative Colitis, Primary Sclerosing Cholangitis (PSC), Primary Biliary Cirrhosis, acute and chronic graft versus host disease (GVHD)).
* Individuals with autoantibodies plus objective evidence of end organ damage related to a cutaneous immune-mediated disease (e.g. psoriasis and mycosis fungoides, etc.) or diseases of the hematopoietic system, liver and the gastrointestinal tract (e.g. aplastic anemia, Crohn's disease, Ulcerative Colitis, Primary Sclerosing Cholangitis (PSC), Primary Biliary Cirrhosis, acute and chronic graft versus host disease (GVHD)).
* Individuals with a history of serious infection within the last 6 months.
* Individuals with tuberculosis, HIV, or hepatitis B, or C.
* Patients unable to provide consent
* Incarcerated individuals

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will use topical imiquimod as standard of care and who are without immune-mediated systemic disease
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Immune response | 5 years
  RNA sequencing of patients to gauge immune response as measured by expression of key inflammatory cytokines related to TLR7 response generated by imiquimod.

SECONDARY OUTCOMES:
Monitoring | 1 year
  Incidence of treatment-related adverse events
Flow cytometry | 3 years
  Flow cytometry measurement of cell populations in patients after imiquimod
Immunohistochemistry | 3 years
  Immunohistochemical staining of patient biopsies using immune cell stains: CD3, CD4, CD8, CD68

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No